CLINICAL TRIAL: NCT06951412
Title: The Effect of Foot Reflexology Massage Applied to Women With Type 2 Diabetes on Neuropathic Pain
Brief Title: The Effect of Foot Reflexology Massage on Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Adile Nese, assoc prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Foot Reflexology
Record Dates: First submitted 2024-06-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
Keywords: Foot massage; Reflexology; Neuropatic pain; Nursing; neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Complementary Therapies

STUDY DESIGN:
Intervention Model Description: At this stage, the patients in the intervention group received a foot reflexology massage by the researcher in the podiatry room of the Endocrinology and Metabolic Diseases polyclinic in a quiet and calm environment for 6 weeks, two sessions per week, for a total of 12 sessions and 30-40 minutes (15-20 minutes for each foot). Data collection forms were filled out for the patients in the control group, but no application was made.
Masking Description: experimental and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The effect of reflexology massage on the average pain score (Experimental): The effect of reflexology massage on neuropathy-related pain score
  Interventions: Other: Foot Reflexology Massage
- The Effect of Foot Reflexology Massage Applied to Women With Type 2 Diabetes on Neuropathic Pain (Experimental): The Effect of Foot Reflexology Massage Applied to Women With Type 2 Diabetes on Neuropathic Pain
  Interventions: Other: Foot Reflexology Massage

INTERVENTIONS:
Other: Foot Reflexology Massage — Reflexology Massage
  Other Names: complementary therapy

SUMMARY:
This study is conducted to measure the effect of foot reflexology massage on neuropathic pain in diabetic patients.Is reflexology foot massage applied to type 2 diabetic patients effective on neuropathic pain?

DETAILED DESCRIPTION:
Controlling pain in individuals with diabetes; It is important for the individual to relax, increase the quality of life, reduce complications and shorten the duration of hospital stay. For this reason, the importance of neuropathic pain and its treatment is increasing in terms of public health. In this study, the effect of foot reflexology massage applied to women with type 2 diabetes on neuropathic pain was measured.

ELIGIBILITY:
Inclusion Criteria:

1. Those diagnosed with type 2 diabetes,
2. Being 18 years or older
3. Individuals who do not have any fractures in the extremities, skin diseases, past wound history, open wounds and unilateral or bilateral amputation, tendonitis in the ankle, active foot ulcer and infection.
4. Those who volunteer to participate in the study,
5. Those who do not have problems with verbal communication,
6. Those who have not been diagnosed with any psychiatric disease.
7. Those with neuropathic pain of 12 points and above according to the LANS score
8. Patients receiving duloxetine drug therapy
9. Those who are not pregnant
10. Patients without peripheral artery disease, deep vein thrombosis and gonatosis will be included in the study. -

Exclusion Criteria:

1. Those who did not agree to participate in the study
2. Those under 18 years of age
3. Individuals with no fractures in the extremities, skin diseases, past wound history, open wounds and unilateral or bilateral amputation, tendonitis in the ankle, active foot ulcers and infections.
4. Those who have problems with verbal communication
5. Those with neuropathic pain below 12 points according to the LANS score
6. Patients receiving treatment other than duloxetine drug therapy
7. Those who are pregnant
8. Those with any psychiatric disorder
9. Patients with peripheral artery disease, deep vein thrombosis and gonatosis will not be included in the study.-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Type 2 Diabetes patients
Enrollment: 65 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
pain score | 6 Weeks
  visual analog scale:VAS: It is a scale scored between 0 and 10 points. A score of 0 indicates that the patient has no pain, and a score of 10 indicates that the patient has unbearable pain. The patient gives a score between 0 and 10 depending on the pain condition.

SECONDARY OUTCOMES:
Four Question Neuropathic Pain Questionnaire | 6 weeks
  This questionnaire consists of a total of 10 items; 7 items are related to the quality of pain (burning, painful cold, electric shocks) and its relationship with abnormal sensations (tingling, pins and needles, numbness, itching), and 3 items are related to the clinical examination of the painful area (touch hypoesthesia, pricking hypoesthesia, tactile allodynia). Each item is scored 1 if the answer is yes and zero if no, with a minimum of zero and a maximum of 10 points. In this assessment, a score of ≥4 out of 10 is considered neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Akarsu, Study Director — Gaziantep University Faculty of Medicine
Locations (1):
- Gaziantep University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paju, W., Yusuf, R., Nurhidayah, J., Fauzi, A., Bata, V. A., & Agustine, U. (2022). The effect of foot massage on peripheral neuropathy in patients with diabetic mellitus: a systematic review. Malaysian Journal of Medicine and Health Sciences, 18(17), 354-362.
- [Background] de Fátima Megda, L., Terra, A. M. S. V., de Matos, J. B., de Melo Taveira, L., Martínez, B. B., de Cássia Pereira, R., ... & Santos, A. T. S. (2020). Immediate effect of foot reflexology in patients with diabetic neuropathy-Randomized Clinical Trial. Revista Neurociências, 28, 1-22.
- [Background] Ibrahim MM, Rizk SMA, The efficacy of foot reflexology on the reduction of peripheral diabetic neuropathic pain. J Nurs Health Sci. 2018; 7(5): 44-55.